CLINICAL TRIAL: NCT01890603
Title: Ambulatory Safety and Quality Program: Improving Management of Individuals With Complex Healthcare Needs Through Health It
Brief Title: Enhancing Complex Care Through an Integrated Care Coordination Information System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Care Management Plus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HS17832
Record Dates: First submitted 2012-01-12; First posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Nurse Based Care Management; Health Information Technology
Keywords: Care coordination, primary care; nurse care management; practice facilitation
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care Coordination Arm (Experimental)
  Interventions: Other: Data collection
- Quality Measure Improvement (Active Comparator)
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data collection — Research involving materials (data, documents, records, or specimens) that have been collected, or will be collected, solely for non-research purposes (such as medical treatment or diagnosis).
  Arms: Care Coordination Arm
Other: Data Collection — Research involving materials (data, documents, records, or specimens) that have been collected, or will be collected, solely for non-research purposes (such as medical treatment or diagnosis).
  Arms: Quality Measure Improvement

SUMMARY:
Cluster randomized controlled trial comparing care coordination incentives to pay for performance (quality measure) incentives in clinics on utilization, cost, quality, and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Six Clinics participating whom Care Management Plus team has worked with before
* Patients belonging to one of these six clinics
* Picked based on an algorithm designed to identify high risk patients.
* Clinic will review potential patients list and issue a survey with consent form

Exclusion Criteria:

* Younger than 18
* Older than 90

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60000 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rate of Utilization | up to 18 months
  Utilization includes Emergency Department visits and hospitalizations for this high risk group.

SECONDARY OUTCOMES:
Patient Satisfaction/Experience | 0, 18 months
  Patient Assessment of Care for Chronic Conditions (PACIC; Consumer Assessment of Healthcare Providers and Systems
Reduce Costs | 0, 12, 18 months
  Costs will be aggregated and compared across groups
Improve quality of care | 0,3,6,9,12,15,18 months
  5 pre-validated quality measures will be aggregated and compared across groups.

CONTACTS AND LOCATIONS:
Overall Officials: David Dorr, MD MS, Principal Investigator — Oregon Health and Science University; Gwenivere Olsen, BS, Study Chair — Oregon Health and Science University; Kelli Radican, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States